CLINICAL TRIAL: NCT05864222
Title: Impact of Aromatherapy on Happiness and Job Satisfaction in Nurses Working in an Academic Health System (AHS)
Brief Title: Aromatherapy and Happiness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-00408
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Happiness
MeSH Terms: interventions — Aromatherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nurses Working in an Academic Health System (AHS) (Experimental): Nurse participants will receive aromatherapy (AT) after baseline measurements. Each day, the participants will pick up AT stickers to wear throughout the day on their staff badges. Participants will receive monthly emails, reminding them to wear the AT every day that they are working.
  Interventions: Other: Aromatherapy

INTERVENTIONS:
Other: Aromatherapy — Elequil Aroma-Tabs are available on all clinical nursing units for staff. Instructions will be provided to participants to place the aroma tab on the back of their badge every workday for the entire duration of their shift. They will wear their badge in whatever position is most comfortable to them for the duration of the study (6 months).
  Other Names: Elequil Aroma-Tabs

SUMMARY:
The purpose of this study is to explore the impact that aromatherapy has on nurses' self-perception of happiness and workplace satisfaction. After completing the informed consent process, participants will complete a demographic survey, the Oxford Happiness Questionnaire (OHQ), and the Nursing Job Satisfaction Survey (NJSS). Aromatherapy (AT), via AT stickers on employee badges, will begin after baseline measurements. OHQ and NJSS will be measured again at 3 months and 6 months of AT. After completion of the intervention, participants will also complete a qualitative survey addressing overall self-reported impact of AT. Analysis will occur after final data is collected.

ELIGIBILITY:
Inclusion Criteria:

1. A Registered Nurse at NYULH
2. Willing to provide an email address of choice
3. Willing to wear an aromatherapy badge sticker during every work shift
4. Not allergic or otherwise sensitive to aromatherapy scent

Exclusion Criteria:

1. Not a Registered Nurse at NYULH
2. Not willing to provide an email of choice
3. Not willing to wear an aromatherapy badge sticker during every work shift
4. Allergic or otherwise sensitive to aromatherapy scent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-02-24 (Actual); Study Completion 2024-02-24 (Actual)

PRIMARY OUTCOMES:
Change in Nursing Job Satisfaction Survey (NJSS) Score | Baseline, Month 6
  23-item assessment of job satisfaction among nurses. Items are ranked on a scale from 0 (strongly disagree) to 4 (strongly agree). The total score ranges from 0 to 92; higher scores indicate greater satisfaction.
Change in Oxford Happiness Questionnaire (OHQ) Score | Baseline, Month 6
  29-item assessment of happiness. Items are ranked on a scale from 1 (strongly disagree) to 6 (strongly agree). Total scores range from 29 to 174; higher scores indicate greater happiness.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen E Zavotsky, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Email is being collected and will be destroyed once data analysis is complete